CLINICAL TRIAL: NCT05967650
Title: Efficacy of Accelerated Versus Standard Regiment of Hepatitis B Virus Vaccine Among Inflammatory Bowel Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Sabry, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HBV vaccines in IBD patients
Record Dates: First submitted 2023-07-08; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Hepatitis B vaccines
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBV vaccination of Inflammatory bowel disease patients with stander regemin (Active Comparator): inflammatory bowel disease patient with negative HBVs AB will be vaccinated with standerd regemin HBV vaccination
  1. st dose zero
  2. nd dose after 2 months
  3. rd dose after 6 months
  Interventions: Biological: standard hepatitis B vaccine
- HBV vaccination of Inflammatory bowel disease patients with accelearetd regemin (Active Comparator): inflammatory bowel disease patient with negative HBVs AB will be vaccinated with standerd regemin HBV vaccination
  1. st dose zero
  2. nd dose after 1months
  3. rd dose after 3 months
  Interventions: Biological: accelerated HBV Vaccine

INTERVENTIONS:
Biological: standard hepatitis B vaccine — IBD patients with negative HBV will be diveded in to two arms first arm vaccinated with standard HBV vaccine regemin( dose 0.2.6)
  Arms: HBV vaccination of Inflammatory bowel disease patients with stander regemin
Biological: accelerated HBV Vaccine — IBD patients with negative HBV will be diveded in to two arms second arm vaccinated with accelerated HBV vaccine regemin( dose 1.2.3)
  Arms: HBV vaccination of Inflammatory bowel disease patients with accelearetd regemin

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract that includes ulcerative colitis (UC) and Crohn's disease (CD) . They mainly affect young populations, altering their quality of life and increasing morbidity, compared to the general population . The etiology and pathogenesis of IBD are still poorly understood.

Inflammatory bowel disease (IBD) patients are at an increased risk of contracting and developing complications from hepatitis B virus (HBV) due to their weakened immune systems and frequent use of immunosuppressive medications. The traditional HBV vaccine regimen requires three doses over six months to achieve full immunity, which can be challenging for IBD patients who may have difficulty adhering to the schedule or may not respond well to the vaccine

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract that includes ulcerative colitis (UC) and Crohn's disease (CD) . They mainly affect young populations, altering their quality of life and increasing morbidity, compared to the general population . The etiology and pathogenesis of IBD are still poorly understood. The pathogenesis of IBD involves genetic factors and environmental factors . In Egypt, the prevalence of IBD has been increasing in recent years.

Patients with inflammatory bowel illnesses are more susceptible to viral infections. In people with IBD, viral infections have emerged as a significant issue. Viral infections are often difficult to identify and have a high morbidity and fatality rate.

The hepatitis B virus is a widespread infection worldwide. HBV is a DNA virus of the Hepadnaviridae family that is a significant cause of morbidity and mortality . Hepatitis B virus (HBV) infection is a global health problem with a continuously increasing burden in developing countries like Egypt.

The prevalence of HBV in Egypt remains a significant public health concern, with a pooled prevalence of 3.67%. However, the introduction of the HBV vaccination program in 1992 has led to a decrease in prevalence among low-risk populations, with a pooled prevalence estimate of 1.93%. This highlights the importance of continued efforts to promote and expand HBV vaccination programs in Egypt.Notably, children under 20 with a history of HBV vaccination in infancy had the lowest prevalence of 0.69%, indicating the effectiveness of HBV vaccination during infancy in providing adequate protection. This underscores the need for increasing vaccination coverage among infants and young children in Egypt.However, the prevalence of HBV in pregnant females was still high among low-risk groups, with a pooled prevalence of 2.9%. This highlights the importance of targeted interventions to prevent mother-to-child transmission of HBV, such as screening pregnant women for HBV and providing antiviral therapy to those who test positive.Overall, while progress has been made in reducing the prevalence of HBV in Egypt, continued efforts are needed to further decrease the burden of this disease and prevent its transmission.

Inflammatory bowel disease (IBD) patients are at an increased risk of contracting and developing complications from hepatitis B virus (HBV) due to their weakened immune systems and frequent use of immunosuppressive medications. The traditional HBV vaccine regimen requires three doses over six months to achieve full immunity, which can be challenging for IBD patients who may have difficulty adhering to the schedule or may not respond well to the vaccine. An accelerated HBV vaccine regimen has been developed that allows for faster immunity with fewer doses, but its efficacy in IBD patients to be investigated.[5]

ELIGIBILITY:
Inclusion Criteria:

* IBD patients with negative HBs Ag and HBsAb less than 10

Exclusion Criteria:

* Patients who refuse enter the study
* Patients who already have HBV infection
* Patients who had HBV vaccine recently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
- efficacy of accelerated HBV vaccine regimen versus standard HBV vaccine regiment among IBD patients already receive treatment | 7 months
  accelearted HBV vaccine will be given at( dose 0 ,1,3) mothns while standard HBV vaccine regemin( dose 0.2.6) efficacy of both regimen assessed by measurement of HBs Ab titre by IU

SECONDARY OUTCOMES:
frequency of IBD patients with negative HBs Ab | 2 months
  All IBD patients at Alraghy hospital will be tested for HBsAg, HBcAb and HBsAb titre by IU

CONTACTS AND LOCATIONS:
Overall Officials: bahaa os taha, Study Chair — Assiut University; lobna ah abdelwahed, Study Director — Assiut University

REFERENCES:
- [Background] Abraham C, Cho JH. Inflammatory bowel disease. N Engl J Med. 2009 Nov 19;361(21):2066-78. doi: 10.1056/NEJMra0804647. No abstract available. PMID 19923578
- [Background] Fabian O, Kamaradova K. Morphology of inflammatory bowel diseases (IBD). Cesk Patol. 2022 Spring;58(1):27-37. PMID 35387455
- [Background] Molodecky NA, Kaplan GG. Environmental risk factors for inflammatory bowel disease. Gastroenterol Hepatol (N Y). 2010 May;6(5):339-46. PMID 20567592
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Kaplan GG, Ng SC. Understanding and Preventing the Global Increase of Inflammatory Bowel Disease. Gastroenterology. 2017 Feb;152(2):313-321.e2. doi: 10.1053/j.gastro.2016.10.020. Epub 2016 Oct 25. PMID 27793607
- [Background] Gholizadeh O, Akbarzadeh S, Moein M, Yasamineh S, Hosseini P, Afkhami H, Amini P, Dadashpour M, Tahavvori A, Eslami M, Hossein Taherian M, Poortahmasebi V. The role of non-coding RNAs in the diagnosis of different stages (HCC, CHB, OBI) of hepatitis B infection. Microb Pathog. 2023 Mar;176:105995. doi: 10.1016/j.micpath.2023.105995. Epub 2023 Jan 18. PMID 36681203
- [Background] Azzam A, Khaled H, Elbohy OA, Mohamed SA, Mohamed SMH, Abdelkader AH, Ezzat AA, Elmowafy AOI, El-Emam OA, Awadalla M, Refaey N, Rizk SMA. Seroprevalence of hepatitis B virus surface antigen (HBsAg) in Egypt (2000-2022): a systematic review with meta-analysis. BMC Infect Dis. 2023 Mar 10;23(1):151. doi: 10.1186/s12879-023-08110-5. PMID 36899311
- [Background] Fernandez Sanchez-Escalonilla S, Esparcia Rodriguez O, Lopez Canto S, Cantero Escribano JM, Molina Cabrero FJ, Gomez-Juarez Sango A, Garcia Guerrero J. [Vaccination against hepatitis B in patients with inflammatory bowel disease: immune response and associated factors.]. Rev Esp Salud Publica. 2022 Feb 18;96:e202202020. Spanish. PMID 35179147
- [Background] Ridola L, Zullo A, Lagana B, Lorenzetti R, Migliore A, Pica R, Picchianti Diamanti A, Gigliucci G, Scolieri P, Bruzzese V. Hepatitis B (HBV) reactivation in patients receiving biologic therapy for chronic inflammatory diseases in clinical practice. Ann Ist Super Sanita. 2021 Jul-Sep;57(3):244-248. doi: 10.4415/ANN_21_03_08. PMID 34554119